CLINICAL TRIAL: NCT03347409
Title: Validation of an ERAS Protocol in Gynecological Surgery: an Italian Randomized Controlled Trial
Brief Title: Validation of an ERAS Protocol in Gynecological Surgery
Acronym: ERASGYNBS001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Federico Ferrari, MD, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP 2722
Record Dates: First submitted 2017-10-27; First posted 2017-11-20 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Surgery; Hysterectomy; Gynecologic Disease; Gynecologic Cancer; Anesthesia
Keywords: ERAS, Fast-track surgery, gynecology
MeSH Terms: conditions — Genital Diseases, Female | interventions — Preoperative Care; Intraoperative Care; Postoperative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Perioperative (SP) care (No Intervention)
- ERAS protocol (Experimental)
  Interventions: Other: Changes in preoperative care; Other: Changes in intraoperative care; Other: Changes in postoperative care

INTERVENTIONS:
Other: Changes in preoperative care — Optimization of relevant medical uncontrolled situations, avoid fasting, avoid bowel preparation, avoid premedications, nutritional assessment, stop smoking, stop alcohol and appropriate counselling
  Arms: ERAS protocol
Other: Changes in intraoperative care — Blended anesthesia is mostly carried out using Total Intra Venous Anesthesia (TIVA) with loco regional analgesia, in particular Thoracic Epidural Anesthesia (TEA) in open surgery and spinal morphine or Transversus Abdominis Plane (TAP) block or quadratus lumborum block for laparoscopic surgical approach, associated to NSAIDs or acetaminophen; control of deep neuromuscular blocking with Train-of-four (TOF) stimulation avoiding residual paralysis. Multimodal prevention of PONV (according to preoperative assessment of Apfel Score) with a combination of multiple antiemetic drugs.
  Arms: ERAS protocol
Other: Changes in postoperative care — Postoperative pain control is obtained with opioid sparing strategies, in order to avoid Post Operative Ileus (POI) and PONV. According to the type of surgery TEA, TAP block , quadratus lumborum block or IT morphine is preferred. Patient is proposed to start drinking clear fluid 4 hours after surgery and to start eating the evening of the surgery, with the introduction of a normal free diet within 24 hours after surgery. It is proposed to chew gum three times daily for at least 15 minutes and eventually to use laxatives to promote a faster bowel function. Early mobilization is started from the evening of surgery.
  Arms: ERAS protocol

SUMMARY:
Validation of ERAS interventional measures in elective gynecological surgery, for benign either malignant pathology.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and <75 years old
* Patients candidated for elective gynecological surgery for benign pathology
* Patients with diagnosis of gynecological neoplasm and candidated for elective gynecological surgery
* Signed consent form
* Karnofsky Performance Status > 70

Exclusion Criteria:

* ASA score > 3
* Contraindication to loco-regional anaesthesia
* Patients with ileus or subocclusive condition prior surgery
* Coagulation disorders
* Organ failure or severe disfunction (heart, renal, pulmonary, hepatic)
* Uncontrolled hypertension (>180/95)
* Alcohol or drug abuser (current or previous)
* Unability to self-care (PFS < 70)
* Comorbidity-Polypharmacy Score > 22
* Psychiatric condition or language barriers
* Planned Intensive Care Recovery

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 166 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-07-14 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Shorter Length Of Hospitalization (LOH) | Up to 4 weeks after surgery
  Total amount of days spent in hospital

SECONDARY OUTCOMES:
Assessment of postoperative pain | At moment 0, 3, 6, 12 and 24 hours after surgery
  NRS scale (from 0 to 10, 0 is no pain, 10 is maximum pain)
Presence/Absence of nausea | At moment 0, 3, 6, 12 and 24 hours after surgery
Presence/Absence of vomiting | At moment 0, 3, 6, 12 and 24 hours after surgery
Anesthesiological complications | Up to 1 weeks after surgery
  Rate measurement
Time to bowel movement | Up to 4 weeks after surgery
  Hours elapsed to event
Time to flatus | Up to 4 weeks after surgery
  Hours elapsed to event
Time to hunger | Up to 4 weeks after surgery
  Hours elapsed to event
Time to drink | Up to 4 weeks after surgery
  Hours elapsed to event
Time to eating | Up to 4 weeks after surgery
  Hours elapsed to event
Time to walking | Up to 4 weeks after surgery
  Hours elapsed to event
Postoperative complications | Up to 9 weeks after surgery
  Rate measurement
Compliance to ERAS protocol | Up to 4 weeks after surgery
  Rate measurement
Validated questionnaires | Administered 24 hours after surgery and up to 4 weeks after surgery
  QoR15

CONTACTS AND LOCATIONS:
Locations (1):
- Federico Ferrari, Brescia, BS, Italy

REFERENCES:
- [Derived] Chau JPC, Liu X, Lo SHS, Chien WT, Hui SK, Choi KC, Zhao J. Perioperative enhanced recovery programmes for women with gynaecological cancers. Cochrane Database Syst Rev. 2022 Mar 15;3(3):CD008239. doi: 10.1002/14651858.CD008239.pub5. PMID 35289396
- [Derived] Ferrari F, Forte S, Sbalzer N, Zizioli V, Mauri M, Maggi C, Sartori E, Odicino F. Validation of an enhanced recovery after surgery protocol in gynecologic surgery: an Italian randomized study. Am J Obstet Gynecol. 2020 Oct;223(4):543.e1-543.e14. doi: 10.1016/j.ajog.2020.07.003. Epub 2020 Jul 8. PMID 32652064